CLINICAL TRIAL: NCT04536181
Title: Comparative Study of 3 or 6 Months Initial Steroid Treatment in Children Under 6 Years of Age With Steroid Sensitive Nephrotic Syndrome：a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Study of Initial Steroid Treatment in Young Children With Nephrotic Syndrome
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSICS
Record Dates: First submitted 2020-08-26; First posted 2020-09-02 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Steroid-Sensitive Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Prednisolone; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 months group (Placebo Comparator): Subjects will receive 12-weeks of placebo following randomization
  Interventions: Drug: Placebo
- 6 months group (Experimental): 12 Weeks of Prednisolone Therapy Subjects will add an additional 12 weeks of Prednisolone to follow pre-randomization standard of care prednisolone.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — 12 weeks prednisolone treatment
  Other Names: prednisone
  Arms: 6 months group
Drug: Placebo — 12 weeks simulated tablets
  Arms: 3 months group

SUMMARY:
This study is a multicentric, prospective, randomized, double blind, placebo controlled trial compared the efficacy of 6 months vs. 3 months of initial prednisolone therapy in decreasing the incidence of FRNS with steroid-sensitive nephrotic syndrome in children age 1 year up to 6 years. Three months tapering prednisolone or placebo are administrated follow by open-label 3 months standard prednisolone therapy.The cumulative incidence of FRNS and adverse events for one year were evaluated in the 3-month and 6-month groups.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic, steroid-sensitive, first episode of nephrotic syndrome
* Age 12 months up to 6 years
* Written informed consent

Exclusion Criteria:

* Nephrotic syndrome known to be secondary to a systemic disorder, e.g., Immunoglobulin A (IgA) nephropathy, systemic lupus erythematosus, Henoch Schonlein purpura, vasculitis, , hepatitis B or Alport syndrome.
* Therapy with prednisolone for prior episodes of nephrotic syndrome
* Persistent estimated glomerular filtration rate (GFR) <75 ml/min/1.73 m2
* Patients who show relapse during the first 3 months of pre-randomization corticosteroid therapy for nephrotic syndrome
* Patients with initial steroid resistance
* Patients who are allergic to glucocorticoids
* The compliance of patients or their guardians is poor

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of frequent relapses of nephrotic syndrome at 12th month after 3 month standard treatment | 12 month period after 3 month standard treatment
  Proportion of patients with frequent relapses at 12th month after 3 month standard treatment.Frequent relapses nephrotic syndrome was defined as two or more relapses within 6 months after completing initial treatment, or four relapses within any period of 12 months, including relapses during initial treatment.

SECONDARY OUTCOMES:
Number of relapses during 12 months follow up after 3 month standard treatment | 12 month period after 3 month standard treatment
  Number of nephrotic syndrome relapses per patient year during the 12-month period after 3 month standard treatment
Time to first relapse (days) | 12 month period after 3 month standard treatment
  Number of days from randomization to occurrence of first relapse
Cumulative prednisolone [or corticosteroid equivalent] received during 12 month period after 3 month standard treatment | 12 month period after 3 month standard treatment
  Total amount of prednisolone [or corticosteroid equivalent] received, as mg/kg/day or mg/m2/day as intervention and for treatment of relapses, during 12 months follow up after 3 month standard treatment
The use of steroid-sparing medications | 12 month period after 3 month standard treatment
  The proportion of patients in each study arm treated with steroid-sparing strategies or medications.it is a binary varibale (1/0). The variable wolud be sette into "1", if the patients use the steroid-sparing medications such as cyclophosphamide, levamisole, mycophenolate mofetil，rituximab and so on.
Adverse events during 12-month period after 3 month standard treatment | 12 month period after 3 month standard treatment
  Number of adverse events experienced, related or unrelated to corticosteroid use
Change in height during 12-month period after 3 month standard treatment | 12 month period after 3 month standard treatment
  The standard deviation scores (SDS) for height will be measured at 12th month and randomization. Change in height is SDS at 12 month minus that of randomization.
Occurrence of steroid-dependent nephrotic syndrome at 12th month after 3 month standard treatment | 12 month period after 3 month standard treatment
  Proportion of patients with steroid-dependent nephrotic syndrome at 12th month after 3 month standard treatment.Steroid-dependent nephrotic syndrome was defined as steroid-sensitive nephrotic syndrome with 2 or more consecutive relapses during tapering or within 14 days of stopping steroids.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Xu, PhD.MD., Principal Investigator — Children's Hospital of Fudan University
Locations (4):
- China (4):
  - Children's hospital of Fudan university, Shanghai, Shanghai Municipality
  - Shanghai Children's Hospital, Shanghai
  - Shanghai Children's Medical Center, Shanghai
  - Xinhua Hospital, Shanghai Jiaotong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No